CLINICAL TRIAL: NCT00069732
Title: Pilot of Two CAM Treatments for Maintenance of Weight Loss
Brief Title: Study of Two Complementary and Alternative Medical Treatments for Maintenance of Weight Loss
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21AT001190-01A1 (NIH); R21AT001190-01A1 (NIH)
Record Dates: First submitted 2003-09-30; First posted 2003-10-03 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2010-02

CONDITIONS: Obesity
Keywords: Overweight; Weight loss maintenance; CAM therapy; Qigong; Acupressure; Traditional Chinese Medicine
MeSH Terms: conditions — Obesity; Overweight | interventions — Qigong

INTERVENTIONS:
Behavioral: qigong
Behavioral: acupressure-TAT

SUMMARY:
The goal of this study is to pilot test in a group of overweight-obese individuals the feasibility and acceptability and indications of efficacy of two CAM treatments, qigong, and acupressure-TAT, for improving long term maintenance of weight loss.

DETAILED DESCRIPTION:
The prevalence of obesity is at epidemic proportions, 60% of US adults are overweight or obese. Obesity contributes to chronic diseases (diabetes, cardiovascular disease [CVD], hypertension, cancer, and osteoarthritis) and to escalating health care costs. Weight loss can have a substantial impact on reducing these conditions. Substantial efforts have been made in developing effective short-term weight loss programs using behavioral treatments. However, long-term maintenance of weight loss continues to be problematic - many individuals regain the weight lost within a year. Innovative intervention options are critically needed to help people successfully maintain weight loss and to fight the obesity epidemic. Complementary and alternative medicine (CAM) approaches-mind-body, energy healing, and Traditional Chinese Medicine (TCM) approaches may hold great promise for helping improve the maintenance of weight loss.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-35 kg/m 2
* Reside in Portland metropolitan area
* Willing to complete the 12-week weight loss program
* Willing to accept random assignment to one of the three maintenance treatment conditions
* Willing to provide informed consent

Exclusion Criteria:

* Medical conditions or treatments that would be contraindicated using a diet & exercise weight loss treatment
* Cancer
* Significant GI disease inappropriate for diet and physical activity intervention
* Diabetes dependent on insulin or oral hypoglycemic medications
* Psychiatric hospitalization in past 2 years
* Conditions that require limitation of physical activity
* Congestive Heart Failure
* Cardiovascular Disease (stroke, MI, CABG, ASCVD)
* Taking weight loss medications currently or within past 6 months
* Previous history of complementary or alternative medicine (CAM) weight loss treatment
* Current acupressure, or Qi Gong, or acupuncture
* Reported consumption of more than 21 alcoholic drinks per week
* Planning to leave the area prior to the end of the program
* Body weight change > 10 pounds in the 6 months prior to Screening visit one
* Pregnant, breast feeding, or planning pregnancy prior to the end of participation
* Current participation in another clinical trial
* Investigator discretion for safety or adherence reasons
* Household member of another CAM WT participant
* Unavailable for group sessions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90

CONTACTS AND LOCATIONS:
Overall Officials: Patricia J Elmer, PhD, Principal Investigator — Center for Health Research, Northwest
Locations (1):
- Center for Health Research, Portland, Oregon, United States